CLINICAL TRIAL: NCT02504151
Title: Cannabidiol Treatment in Patients With Early Psychosis
Acronym: CBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, MD, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1412015000
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cannabidiol, then Placebo (Experimental): The subject will receive treatment with cannabidiol (CBD)(800mg/day) for four weeks, followed by a two week washout period, followed by four weeks of placebo.
  Interventions: Drug: Cannabidiol; Drug: Placebo
- Placebo, then Cannabidiol (Experimental): The subject will receive placebo for four weeks, followed by a two week washout period, followed by four weeks of treatment with cannabidiol (CBD)(800mg/day).
  Interventions: Drug: Cannabidiol; Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol
  Other Names: CBD
Drug: Placebo

SUMMARY:
Cannabidiol (CBD) is a component of herbal cannabis that is present in varying concentrations in cannabis extracts. CBD has been shown to produce central effects including hypnotic, anticonvulsive, anxiolytic and neuroprotective effects.The investigators hypothesize that treatment with CBD will result in: 1) Improvement evidenced by a reduction in scores on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS), 2) Improvement evidenced by a reduction in the Clinical Global Impression of Severity scale (CGI); Secondary Hypothesis: 1) Greater improvement in functioning as measured on the "Patient Assessment of Own Functioning Inventory: (PAOFI) and the Quality of Life Scale (QLS) In this 2 period cross over design, subjects will be randomized in a 1:1 ratio to receive either: Order 1: CBD (Period 1) followed by placebo (Period 2) or Order 2: Placebo (Period 1) followed by CBD (Period 2) under double-blind conditions. The 2 study periods will be separated by a washout of at least 2 weeks. During each period subjects will receive study medications (CBD [total 800mg/day] or placebo) for a period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Primary psychotic disorder
* Ages 18-65 (inclusive)

Exclusion Criteria:

* Current significant medical condition or other comorbidities
* Current substance depdendence
* Women who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- Cannabidiol, Then Placebo: The subject will receive treatment with Cannabidiol (CBD) (800 mg/day) for four weeks, followed by a two week washout period, followed by four weeks of placebo.
  Period 1: CBD, 800 mg/day Period 2: Placebo
- Placebo, Then Cannabidiol: The subject will receive placebo for four weeks, followed by a 2 week washout period, followed by four weeks of treatment with Cannabidiol (CBD) (800 mg/day).
  Period 1: Placebo Period 2: CBD, 800 mg/day
Period: First Intervention (4 Weeks)
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 8 | 10
Completed | 7 | 9
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1
Period: Washout (2 Weeks)
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 7 | 9
Completed | 6 | 9
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 6 | 9
Completed | 4 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Full Range); unit: years] | 22.875 [19 to 26] | 26.1 [22 to 29] | 25 [19 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 1 | 3 | 4
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS) Over Time
Description: The Positive and Negative Syndrome Scale is a 30-item scale to assess both the positive and negative symptom symptoms of schizophrenia. The range total score is 30-210. An improvement in symptoms is reflected by a lower score.
Time Frame: Completed each time subject is seen over 10 weeks (screening, period 1 baseline, period 1 week 1, period 1 week 2, period 1 week 3, period 1 week 4, period 2 baseline, period 2 week 1, period 2 week 2, period 2 week 3, period 2 week 4)
Population: The number analyzed in one or more rows differ from the overall number analyzed to reflect the number of participants who completed the scale during each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Number analyzed (Participants) | 8 | 10
score on a scale
  Baseline period 1 | 81.3 (2.8) | 84.0 (2.3)
  Week 1 period 1 | 78.3 (2.8) | 75.3 (2.3)
  Week 2 period 1 | 81.4 (2.8) | 73.9 (2.3)
  Week 3 period 1 | 79.6 (2.8) | 70.6 (2.4)
  Week 4 period 1 | 72.0 (2.8) | 69.0 (2.0)
  Baseline period 2: number analyzed (Participants) | 6 | 9
  Baseline period 2 | 71.9 (3.4) | 68.5 (2.4)
  Week 1 period 2: number analyzed (Participants) | 6 | 9
  Week 1 period 2 | 75.2 (3.4) | 67.6 (2.5)
  Week 2 period 2: number analyzed (Participants) | 6 | 9
  Week 2 period 2 | 72.7 (3.4) | 70.1 (2.5)
  Week 3 period 2: number analyzed (Participants) | 6 | 9
  Week 3 period 2 | 73.2 (3.4) | 69.7 (2.6)
  Week 4 period 2: number analyzed (Participants) | 6 | 9
  Week 4 period 2 | 72.4 (3.4) | 66.9 (2.6)
Statistical Analysis 1: Comparison: Cannabidiol, Then Placebo vs Placebo, Then Cannabidiol; The p value is based on the interaction of treatment and time; Test type: Superiority; p = 0.08, Mixed Models Analysis; Linear mixed models was used with treatment, time and time*treatment interaction in the model; Mean Difference (Net) = -.284, 95% CI 2-sided [-2.28 to 1.71], Standard Error of Mean 1.01 — This is the estimated difference between treatment groups (cbd - placebo)

2. Primary Outcome: Clinical Global Impression of Severity Scale Over Time
Description: Clinical Global Impression of Severity Scale score is a global rating of improvement scale, which requires subjects to rate their degree of improvement on a 7-point scale. The total range score is 1-7. A reduction in scores indicates improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Number analyzed (Participants) | 8 | 10
score on a scale
  Baseline period 1 | 4.1 (0.2) | 4.2 (0.2)
  Week 1 period 1 | 4.1 (0.2) | 4.2 (0.2)
  Week 2 period 1 | 4.4 (0.2) | 4.2 (0.2)
  Week 3 period 1 | 4.4 (0.2) | 4.4 (0.2)
  Week 4 period 1 | 4.3 (0.2) | 4.4 (0.2)
  Baseline period 2: number analyzed (Participants) | 6 | 9
  Baseline period 2 | 4.3 (0.2) | 4.3 (0.2)
  Week 1 period 2: number analyzed (Participants) | 6 | 9
  Week 1 period 2 | 4.3 (0.2) | 4.0 (0.2)
  Week 2 period 2: number analyzed (Participants) | 6 | 9
  Week 2 period 2 | 4.3 (0.2) | 4.4 (0.2)
  Week 3 period 2: number analyzed (Participants) | 6 | 9
  Week 3 period 2 | 4.3 (0.2) | 4.2 (0.2)
  Week 4 period 2: number analyzed (Participants) | 6 | 9
  Week 4 period 2 | 4.3 (0.2) | 4.2 (0.2)
Statistical Analysis 1: Comparison: Cannabidiol, Then Placebo vs Placebo, Then Cannabidiol; The p value is based on the interaction of treatment and time; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.12 to 0.07], Standard Error of Mean 0.05 — This is the estimated difference between treatment groups (cbd - placebo)

3. Secondary Outcome: Patient Assessment of Own Functioning Inventory (PAOFI) Over Time
Description: The PAOFI measures subjects' perceptions of functioning when performing everyday tasks and activities that reflect cognitive strengths and weaknesses. Subjects rate each item on a scale ranging from 0 (almost never) to 5 (almost always). The total score is the sum of the responses to each item (score of 0 to 160). High scores on the PAOFI subscales are indicative of poor perceived cognitive functioning. This scale was modified to remove 3 items- so the highest possible score is 145 for this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Number analyzed (Participants) | 8 | 10
score on a scale
  Baseline period 1 | 90.1 (11.3) | 85.1 (9.4)
  Week 1 period 1 | 85.3 (11.3) | 87.5 (9.4)
  Week 2 period 1 | 95.3 (11.3) | 74.9 (9.4)
  Week 3 period 1 | 93.0 (11.3) | 89.9 (9.4)
  Week 4 period 1 | 95.6 (11.3) | 89.0 (9.6)
  Baseline period 2: number analyzed (Participants) | 6 | 9
  Baseline period 2 | 105.4 (12.2) | 87.3 (9.6)
  Week 1 period 2: number analyzed (Participants) | 6 | 9
  Week 1 period 2 | 108.4 (12.2) | 88.5 (9.7)
  Week 2 period 2: number analyzed (Participants) | 6 | 9
  Week 2 period 2 | 104.7 (12.2) | 90.7 (9.7)
  Week 3 period 2: number analyzed (Participants) | 6 | 9
  Week 3 period 2 | 105.2 (12.2) | 86.3 (9.9)
  Week 4 period 2: number analyzed (Participants) | 6 | 9
  Week 4 period 2 | 107.2 (12.2) | 95.6 (9.9)
Statistical Analysis 1: Comparison: Cannabidiol, Then Placebo vs Placebo, Then Cannabidiol; The p value is based on the interaction of treatment and time; Test type: Superiority; p = 0.485, Mixed Models Analysis; Mean Difference (Net) = -4.97, 95% CI 2-sided [-9.87 to -0.06], Standard Error of Mean 2.47 — This is the estimated difference between treatment groups (cbd - placebo)

4. Secondary Outcome: Quality of Life Scale (QLS) Over Time
Description: The Quality of Life Scale (QLS) is a 21-item scale rated from a semi structured interview, each item is rated 0-6. The specific descriptors vary among items, but the high end of the scales (scores of 5 and 6) reflects normal or unimpaired functioning, and the low end of the scales (scores of 0 and 1) reflects severe impairment of the function in question. A highest score of 126 would indicate unimpaired functioning.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Number analyzed (Participants) | 8 | 10
score on a scale
  Baseline period 1 | 70.4 (7.7) | 72.9 (6.4)
  Week 1 period 1 | 73.4 (7.7) | 74.9 (6.4)
  Week 2 period 1 | 69.9 (7.7) | 67.1 (6.4)
  Week 3 period 1 | 69.0 (7.7) | 71.1 (6.4)
  Week 4 period 1 | 72.3 (7.7) | 70.7 (6.5)
  Baseline period 2: number analyzed (Participants) | 6 | 9
  Baseline period 2 | 68.6 (8.6) | 73.3 (6.5)
  Week 1 period 2: number analyzed (Participants) | 6 | 9
  Week 1 period 2 | 68.6 (8.6) | 76.7 (6.7)
  Week 2 period 2: number analyzed (Participants) | 6 | 9
  Week 2 period 2 | 70.1 (8.6) | 77.6 (6.7)
  Week 3 period 2: number analyzed (Participants) | 6 | 9
  Week 3 period 2 | 66.3 (8.6) | 78.1 (6.8)
  Week 4 period 2: number analyzed (Participants) | 6 | 9
  Week 4 period 2 | 71.8 (8.6) | 82.7 (6.8)
Statistical Analysis 1: Comparison: Cannabidiol, Then Placebo vs Placebo, Then Cannabidiol; The p value is based on the interaction of treatment and time; Test type: Superiority; p = 0.994, Mixed Models Analysis; Mean Difference (Net) = 4.13, 95% CI 2-sided [0.07 to 8.19], Standard Error of Mean 2.05 — This is the estimated difference between treatment groups (cbd - placebo)

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were reported at each visit through the duration of the study at 8 weeks.
Description: AEs were collected by randomization arm, not by intervention method (order in the crossover).
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/10
Other Adverse Events (participants affected / at risk) | 5/8 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol, Then Placebo (N=8) | Placebo, Then Cannabidiol (N=10)
Hospitalization (Psychiatric disorders) | 2 (2) | 0 (0) — Subject experienced a worsening in symptoms
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol, Then Placebo (N=8) | Placebo, Then Cannabidiol (N=10)
Dry mouth (General disorders) | 1 (1) | 2 (2)
Depressed mood, racing thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
ER Visit (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Subject went to ER because of pain from her IUD - was sent home same day and instructed to make an appointment with her OB/GYN
Tension headache (General disorders) | 1 (1) | 0 (0)
Migraine (General disorders) | 1 (2) | 0 (0)
Sedation (General disorders) | 1 (1) | 0 (0) — Subject was in wash out period, not taking the study medication
Scratchy throat and cold symptoms (General disorders) | 0 (0) | 1 (1)
Stye in left eye (Eye disorders) | 0 (0) | 1 (1)
Right shin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Occurred after using a new body wash
Increased itchiness of rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Caused by previous condition (COPD)
Increased tiredness (General disorders) | 0 (0) | 1 (1)
Pain in right forearm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Veisalgia (General disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
High blood pressure/hospitalization (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Relapse to PCP, LSD, and opiate use (General disorders) | 1 (1) | 0 (0)
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash around tattoo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleeplessness (General disorders) | 0 (0) | 1 (1)
Pulled leg muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea/gas
Tingling and numbness on right side to body and face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swollen left foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening of symptoms and more negative affect (Psychiatric disorders) | 0 (0) | 1 (1)
Flu (General disorders) | 1 (1) | 0 (0)
Sinusitis (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02504151/Prot_SAP_000.pdf